CLINICAL TRIAL: NCT03658707
Title: Validity and Reliability of the Turkish Version of the Functional Shoulder Score in Patients With Subacromial Impingement Syndrome
Brief Title: Validity and Reliability of the Turkish Version of the Functional Shoulder Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Karabay, Principal investigator, Izmir Katip Celebi University
Other Study IDs: 3864-GOA
Record Dates: First submitted 2018-09-02; First posted 2018-09-05 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Functional shoulder score; questionnaire; subacromial impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Shoulder questionnaire

SUMMARY:
The aim of this study is to determine the validity and reliability of the Turkish version of the Functional Shoulder Score in Turkish patients with subacromial impingement syndrome (SIS).

DETAILED DESCRIPTION:
The original form of the Functional Shoulder Score will be translated into Turkish by two Turkish mother tongue translators who also speak English in advanced level. Then these translations will be combined into one translation and translated back to English. The pre-final version will be composed and tested on a group of patients with SIS. If necessary, readjustments will be made, and the validity of the final version will be investigated in 116 patients with SIS. Additionally, for the test-retest reliability, 59 patients will fill out the questionnaire again after 3-7 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subacromial impingement syndrome (Michener et al, 2009)
* To read and understand Turkish

Exclusion Criteria:

* 50% limitation of passive shoulder range of motion in ≥ 2 planes of motion
* Glenohumeral instability
* Fracture or surgery history in the shoulder
* Another diagnosis that may affect shoulder function (frozen shoulder, primary shoulder arthritis, inflammatory/ neoplastic/neurological conditions, cervical spine induced pain)
* Systemic musculoskeletal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subacromial impingement syndrome from the outpatient clinic of the Dokuz Eylul University, Faculty of Medicine, Department of Orthopedics and Traumatology.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Functional Shoulder Score | Baseline - within 3-7 days after the baseline
  The questionnaire includes 11 items: One is about shoulder pain intensity and 10 is about the shoulder function. The minimum score is 0 (worst) and the maximum score is 100 (best).

SECONDARY OUTCOMES:
Modified Constant Murley Shoulder Score | Baseline
  100 points total score of this score consists of 15 points of pain, 20 points of daily activities, 40 points of the active range of motion, and 25 points of strength. The minimum score is 0 (worst) and the maximum score is 100 (best).
American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form | Baseline
  The patient self-evaluation questionnaire includes 11 item; one is about shoulder pain intensity and 10 are about the shoulder function.The minimum score is 0 (worst) and the maximum score is 100 (best).
Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) | Baseline
  The disability level of the upper extremity is determined by 30 questions; 21 questions are about physical function, 3 questions are about social/role function and 6 questions are about the symptoms of the patient. The minimum score is 0 (best) and the maximum score is 100 (worst).
Western Ontario Rotator Cuff (WORC) index | Baseline
  The disease-specific questionnaire includes 21 items, 4 about physical symptoms, 4 about sport/recreation, 4 about work, 4 about lifestyle and 4 about emotions. The minimum score is 0 (worst) and the maximum score is 100 (best).
Global rating scale | Baseline
  The global shoulder function is graded between 0 (no use) and 10 (normal function) on a scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESILYAPRAK, PhD, Study Director — Dokuz Eylul University; Halime Ezgi TURKSAN, Study Chair — Dokuz Eylul University; Mehmet ERDURAN, MD, Study Chair — Dokuz Eylul University; Damla KARABAY, MSc, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No